CLINICAL TRIAL: NCT03473717
Title: Comparaison de la Douleur Lors de la Pose Des DIU et SIU Entre la méthode Classique et la méthode Directe
Brief Title: Comparison of Pain Level During Intrauterine Device (IUD) Insertion Between Conventional and Direct Method
Acronym: KIDDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-ECO Clinical trial unit on health Economics, Hotel-Dieu Hospital (Unknown); EA 7334 Patient-Centered Outcomes Research, University Paris-Diderot (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HAO 180104
Record Dates: First submitted 2018-03-09; First posted 2018-03-22 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-02

CONDITIONS: IUD Insertion
Keywords: pain; Intrauterine device (IUD); Intrauterine system (IUS); Patient-Reported Outcome
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- classic method group (Active Comparator): IUD/IUS insertion will be done using the conventional method
  Interventions: Device: classic method
- direct method group (Active Comparator): IUD/IUS insertion will be done using the direct method
  Interventions: Device: direct method

INTERVENTIONS:
Device: classic method — * Put the Pozzi forceps to draw the uterus by the cervix to horizontalize it and align uterine cavity in the direct axis of cervix.
  * Insert the hysterometer to measure the uterus depth.
  * Locate the uterine depth on the inserter tube.
  Arms: classic method group
Device: direct method — * Place the ring on the inserter tube 3 to 4 cm from the end as a marker.
  * Insert the tube into the cervix until you feel the passage of the internal orifice of the cervix or until the ring is in contact with the external orifice of the cervix, the tube does not enter the uterine cavity
  Arms: direct method group

SUMMARY:
The so-called "direct" method of intrauterine device (IUD) and intraintuerine system (IUS) insertion is increasingly used. A study has shown that it is technically simpler and assumes less painful than the classic pose.

It seems interesting to compare the pain felt by the patients during IUD / IUS insertion in these two methods of placement and also to confirm that there is no more malposition with the direct method.

DETAILED DESCRIPTION:
The classic method uses: a Pozzi for pulling the uterus to horizontalize it and a hysterometer to visualize the axis of the uterus and to measure the distance between the external orifice of the cervix and the uterine fundus in order to deploy the IUD / IUS.

In the so-called direct technique, the operator does not measure the depth of the uterus thanks to a hysterometer and does not draw the cervix with a Pozzi forceps, the IUD / IUS is deployed as soon as the orifice passes. inside the cervix and the inserter tube does not enter the uterine cavity. With this method the Pozzi forceps is only used as a second line, especially in case of a fleeing neck.

ELIGIBILITY:
Inclusion Criteria:

* The study population will concern all women aged 18 to 50 who want IUD or SIU contraception regardless of whether they are nulliparous, primiparous or pluriparous, whether or not they have had an IUD or IUS.
* Having signed informed consent.
* Being affiliated to a social security scheme (excluding AME)

Exclusion Criteria:

* Can not express their consent
* Not mastering French
* With a contraindication to the chosen IUD or IUS.
* Having had local anesthesia of the cervix (in case of Voluntary Interruption of Pregnancy on the day of insertion)
* Having received analgesic treatment within four hours
* Patient without social security
* No consent of the patient
* Minor patient

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — the study concerns women who want IUD or SIU contraception
Enrollment: 158 (Estimated)
Dates: Start 2018-03-30 (Estimated); Primary Completion 2018-10-15 (Estimated); Study Completion 2019-03-15 (Estimated)

PRIMARY OUTCOMES:
Pain level during the insertion of IUD or IUS | during the procedure of IUD/IUS insertion
  Evaluation endpoint is pain felt by the patient during insertion of the IUD or IUS by a 0-100 mm standard visual analog scale (VAS)

SECONDARY OUTCOMES:
IUD or SIU localization | Ultrasound control performed six to ten weeks after the pose.
  localization of IUD/IUS will be controlled by a pelvic ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Soulat, Principal Investigator — CIVG Hôpital Louis Mourier, AP-HP
Locations (10):
- France (10):
  - CIVG Hôpital Avicenne, Bobigny
  - CIVG Hôpital Louis Mourier, Colombes
  - Liberal Cabinet Midwife, Courbevoie
  - Liberal Cabinet Midwife, Fontenay-sous-Bois
  - Centre de Santé Gatineau Saillant, Gennevilliers
  - CPEF, Gennevilliers
  - Medical Office Gynecology, Paris
  - Hôpital Trousseau, Paris
  - ACSBE-La place santé, Saint-Denis
  - Medical Practice General Practice, Villeneuve-la-Garenne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Golightly E, Gebbie AE. Low-lying or malpositioned intrauterine devices and systems. J Fam Plann Reprod Health Care. 2014 Apr;40(2):108-12. doi: 10.1136/jfprhc-2013-100684. Epub 2014 Jan 6. PMID 24395060
- [Background] Heinemann K, Reed S, Moehner S, Minh TD. Risk of uterine perforation with levonorgestrel-releasing and copper intrauterine devices in the European Active Surveillance Study on Intrauterine Devices. Contraception. 2015 Apr;91(4):274-9. doi: 10.1016/j.contraception.2015.01.007. Epub 2015 Jan 16. PMID 25601352
- [Background] Braaten KP, Benson CB, Maurer R, Goldberg AB. Malpositioned intrauterine contraceptive devices: risk factors, outcomes, and future pregnancies. Obstet Gynecol. 2011 Nov;118(5):1014-1020. doi: 10.1097/AOG.0b013e3182316308. PMID 22015868
- [Background] Teal SB, Romer SE. Awareness of long-acting reversible contraception among teens and young adults. J Adolesc Health. 2013 Apr;52(4 Suppl):S35-9. doi: 10.1016/j.jadohealth.2013.01.013. PMID 23535055
- See also: Related Info — http://bibnum.univ-lyon1.fr/nuxeo/nxbigfile/default/5e9cfad7-7c46-4b51-b737-7cc469e500a9/blobholder:0/Msfb_2014_PETIT_Marion.pdf